CLINICAL TRIAL: NCT03359837
Title: A 26-Week, Multi-Center, Open-label, Randomized, Parallel-group Study to Evaluate the Efficacy and Safety of Two Treatment Regimens in Patients With Type 2 Diabetes After Short-Term Intensive Insulin Therapy: Basal Insulin Based Treatment (With Prandial OADs Combination) Versus Twice-daily Premixed Insulin
Brief Title: Comparison of Two Treatment Regimens in Patients With Type 2 Diabetes After Short-term Intensive Insulin Therapy
Acronym: SWITCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTUL07194; U1111-1186-3400 (Other: UTN)
Record Dates: First submitted 2017-11-21; First posted 2017-12-02 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; insulin glulisine; insulin aspart, insulin aspart protamine drug combination 30:70; repaglinide; Acarbose; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glargine based therapy (Experimental): Once daily glargine plus prandial oral anti-hyperglycemic drugs
  Interventions: Drug: INSULIN GLARGINE (HOE901); Drug: Insulin Glulisine; Drug: Repaglinide; Drug: Acarbose
- Premixed insulin (Active Comparator): Twice daily premixed insulin
  Interventions: Drug: Biphasic insulin aspart 30; Drug: Metformin

INTERVENTIONS:
Drug: INSULIN GLARGINE (HOE901) — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous injection
  Other Names: Lantus
  Arms: Glargine based therapy
Drug: Insulin Glulisine — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous injection
  Other Names: Apidra
  Arms: Glargine based therapy
Drug: Biphasic insulin aspart 30 — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous injection
  Other Names: Novolog Mix70/30
  Arms: Premixed insulin
Drug: Repaglinide — Pharmaceutical form: tablet
  Route of administration: oral administration
  Other Names: NovoNorm
  Arms: Glargine based therapy
Drug: Acarbose — Pharmaceutical form: tablet
  Route of administration: oral administration
  Other Names: Glucobay
  Arms: Glargine based therapy
Drug: Metformin — Pharmaceutical form: tablet or capsule
  Route of administration: oral administration
  Arms: Premixed insulin

SUMMARY:
Primary Objective:

To test the hypothesis that basal insulin based treatment (G+) is noninferior to twice-daily premixed insulin (PM-2) in term of hemoglobin A1c (glycosylated hemoglobin, HbA1c) reduction from baseline to end of study. The test for superiority can be done if noninferiority is achieved.

Secondary Objectives:

* To assess efficacy in terms of percentage of patients achieving HbA1c <7% and HbA1c <7% without hypoglycemia.
* To assess efficacy in terms of percentage of patients achieving fasting plasma glucose (FPG) <7 mmol/L and FPG <7 mmol/L without hypoglycemia.
* To assess safety in term of occurrence of moderate/severe hypoglycemia.
* To assess daily blood glucose (BG) variation.
* To assess patient satisfaction.

DETAILED DESCRIPTION:
The duration of study is approximately 21 months. Each patient will be followed for approximately 27 weeks from screening visit to end-of-study

ELIGIBILITY:
Inclusion criteria :

* Patients with age between 18 and 70 years.
* Hemoglobin A1c>7.5%, and ≤11%.
* Fasting plasma glucose >7 mmol/L.
* Fasting C peptide >1 ng/mL.
* Type 2 diabetes (T2DM) patients with diabetes diagnosis between 2 and 10 years (World Health Organization 1999 T2DM diagnose criteria).
* Continuous treatment with stable doses of metformin (≥1 g/day) and 1 oral antihyperglycemic drug (at least half maximum dose) for more than 3 months prior to screening.
* Body mass index ≥21 kg/m2, and <40 kg/m2.

Exclusion criteria:

* More than 7 consecutive days of insulin treatment within the 12 months except for acute disease or surgery.
* Diabetes other than T2DM (e.g. type 1 diabetes, diabetes secondary to pancreatic disorders, drug or chemical agent intake).
* History of hypoglycemia unawareness or recurrent hypoglycemia or severe hypoglycemia within the past 12 months.
* History of sensitivity to the study drugs or to drugs with a similar chemical structure.
* Pregnancy or planned pregnancy or current lactation (women of childbearing potential must have a negative pregnancy test at study entry and a medically approved contraception method).
* Acute diabetic complications (diabetic ketoacidosis, lactic acidosis, hyperosmolar nonketotic diabetic coma) within the past 12 months.
* Significant diabetic complications and serious disease, e.g., symptomatic autonomic neuropathy, gastroparesis, unstable angina or active proliferative retinopathy.
* Acute infections which may affect BG control within the past 4 weeks.
* Active liver disease, alanine transaminase (ALT) and/or aspartate aminotransferase (AST) greater than two times the upper limit of the reference range at screening.
* Impaired renal function, defined as but not limited to, serum creatinine levels ≥1.5 mg/dL (132 μmol/L) for males and ≥1.4 mg/dL (123 μmol/L) for females or presence of macroproteinuria (>2 g/day).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin A1c (HbA1c) | Baseline to Week 24
  Change in HbA1c from baseline to week 24

SECONDARY OUTCOMES:
Patients with fasting plasma glucose (FPG) <6.1 mmol/L | At Week 12 and Week 24
  Percentage of patients with FPG <6.1 mmol/L at week 12 and week 24
Patients with FPG <6.1 mmol/L without hypoglycemia | At Week 12 and Week 24
  Percentage of patients with FPG <6.1 mmol/L without hypoglycemia at week 12 and week 24
Patients with FPG <7 mmol/L | At Week 12 and Week 24
  Percentage of patients with FPG <7 mmol/L at week 12 and week 2
Patients with FPG <7 mmol/L without hypoglycemia | At Week 12 and Week 24
  Percentage of patients with FPG <7 mmol/L without hypoglycemia at week 12 and week 24
Patients with HbA1c <7% | At Week 12 and Week 24
  Percentage of patients with HbA1c <7% at week 12 and week 24
Patients with HbA1c <7% without hypoglycemia | At Week 12 and Week 24
  Percentage of patients with HbA1c <7% without hypoglycemia at week 12 and week 24
Hypoglycemic events | Baseline to Week 24
  Incidence of hypoglycemia during treatment period
Change in FPG | Baseline to Week 24
  Change in FPG from baseline to week 24
Change in body weight | Baseline to Week 24
  Change in body weight from baseline to week 24
Insulin dose | At Week 24
  Total daily insulin dose at week 24
Daily BG variation at week 24 | At Week 24
  Daily blood glucose (BG) variation at week 24
European quality of life - 5 dimensions (EQ-5D) | Baseline to Week 24
  Change in quality of life scores from baseline to week 24 on 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is measured at 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problem.
Subgroup analysis | At week 24
  Subgroup analysis of control rate of HbA1c <7% according to duration of diabetes, oral anti-hyperglycemic drug(OAD) treatment and HbA1c at screening, FPG, post prandial glucose(PPG) excursion and C peptide at the beginning of run-in period, insulin dose at end of run-in period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- CHINA, China, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Liu J, Jiang X, Xu B, Wang G, Cui N, Zhang X, Liu J, Mu Y, Guo L. Efficacy and Safety of Basal Insulin-Based Treatment Versus Twice-Daily Premixed Insulin After Short-Term Intensive Insulin Therapy in Patients with Type 2 Diabetes Mellitus in China: Study Protocol for a Randomized Controlled Trial (BEYOND V). Adv Ther. 2020 Apr;37(4):1675-1687. doi: 10.1007/s12325-020-01265-6. Epub 2020 Mar 4. PMID 32130661